CLINICAL TRIAL: NCT03169374
Title: Virtual Reality for Anxiety Management in Mechanically Vented Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00000220
Record Dates: First submitted 2017-05-17; First posted 2017-05-30 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Situational Anxiety
Keywords: Virtual Reality; Mechanical Ventilation; Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual Reality Technology (Experimental): Virtual Reality Therapy
  Interventions: Device: Virtual Reality Technology

INTERVENTIONS:
Device: Virtual Reality Technology — Patients in this arm will participate in virtual reality sessions planned for 5 minutes at a time, during which they are shown relaxing virtual environments.

SUMMARY:
The purpose of this study is to investigate the safety and feasibility of virtual reality for anxiety treatment in mechanically ventilated patients.

DETAILED DESCRIPTION:
Mechanically ventilated patients (those on a breathing machine) often experience heightened levels of anxiety and discomfort. This is usually treated by using sedative medications, however these drugs often have unintended side effects. This study will investigate the safety and feasibility of using relaxing virtual reality environments for reduction of anxiety in mechanically ventilated patients.

ELIGIBILITY:
Inclusion Criteria:

Age: 18 years or older

1. Mechanically ventilated; defined as having an endotracheal tube or tracheostomy and requiring continuous support from a mechanical ventilator.
2. Able to spontaneously maintain a state of wakefulness and alertness and able to follow commands
3. Able to communicate with research staff; defined as writing or head nods/shakes

Exclusion Criteria:

1. Delirious; defined as positive on the Confusion Assessment Method for the ICU (CAM-ICU +)
2. Expected to be liberated from ventilator within 12 hours of potential enrollment
3. Existence of skull injury or recent surgery (craniectomy) which precludes safely wearing VR visor
4. Impaired ability to see or hear, as determined by study investigator
5. Ventilator settings with positive end expiratory pressure (PEEP) greater than 10
6. Inability to be safely removed from physical restraints for VR (virtual reality) sessions
7. Chronic ventilator dependence prior to the present hospitalization
8. Lacking capacity to consent for one's self
9. Known difficult airway; based on review of intubation note
10. Tracheostomy performed within last seven days
11. Pre-existing symptoms overlapping with major symptoms of cyber-sickness: Headache, Vertigo (dizziness), Ataxia (tremor with movement), Nausea, Vomiting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of safety events | Immediately following treatment session
  Occurrence rate of safety events, defined as cardiac arrhythmias, hypotension, hypertension, oxygen desaturation, falls to the floor, or unintentional removal of a medical tube or device.

SECONDARY OUTCOMES:
Change in anxiety level during virtual reality treatment | Immediately following treatment session
  Change in anxiety score from pre- to post-virtual reality treatment using a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: David Wacker, M.D., Principal Investigator — University of Minnesota
Locations (1):
- Fairview Southdale Hospital, Edina, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No